CLINICAL TRIAL: NCT00040378
Title: Prevention of Alzheimer's Disease by Vitamin E and Selenium (PREADVISE)
Status: Completed | Type: Observational
Sponsor: Frederick Schmitt (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Frederick Schmitt, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: IA0033; 5R01AG019241 (NIH); NCT00780689 (obsolete NCT alias)
Record Dates: First submitted 2002-06-25; First posted 2002-06-27 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Vitamin E; Selenium
MeSH Terms: conditions — Alzheimer Disease | interventions — Vitamin E; Selenium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Combination therapy: vitamin E (alphatocopherol) and selenium
  Interventions: Drug: alphatocopherol; Drug: Selenium
- Vitamin E only: vitamine E (alphatocopherol) and placebo
  Interventions: Drug: alphatocopherol; Drug: Placebo replacement for Selenium
- Selenium only: selenium and placebo (Placebo replacement for vitamin E)
  Interventions: Drug: Selenium; Drug: Placebo replacement for vitamin E
- Placebo: placebo (Placebo replacement for vitamin E) and placebo (Placebo replacement for selenium)
  Interventions: Drug: Placebo replacement for vitamin E; Drug: Placebo replacement for Selenium

INTERVENTIONS:
Drug: alphatocopherol — 400 IU daily
  Other Names: Vitamin E
  Groups: Combination therapy; Vitamin E only
Drug: Selenium — 200mcg daily
  Groups: Combination therapy; Selenium only
Drug: Placebo replacement for vitamin E — 1 placebo pill daily
  Groups: Placebo; Selenium only
Drug: Placebo replacement for Selenium — 1 placebo pill daily
  Groups: Placebo; Vitamin E only

SUMMARY:
The Prevention of Alzheimer's Disease by Vitamin E and Selenium (PREADVISE) prevention trial is an important addition to the Selenium and Vitamin E Cancer Prevention Trial (SELECT). As a prevention trial, PREADVISE is trying to find out if taking selenium and/or Vitamin E supplements can help to prevent memory loss and dementia such as Alzheimer's disease.

DETAILED DESCRIPTION:
Studies show that increased oxidative stress (from excess free radicals) may damage brain cells and is linked with Alzheimer's disease (AD). Many studies show increased oxidation of brain lipids (fats), proteins, carbohydrates (sugars) and DNA in AD. Although the causes of AD are not known, it is believed that oxidative stress is part of what damages brain cells in AD and probably other brain diseases. Animal and tissue culture studies of vitamin E and selenium suggest that they can protect brain cells from damage. This research study is being done to see how safe and effective vitamin E and selenium may be in preventing AD and other brain illnesses. These illnesses are more common in people over the age of 60 to 65. A potential benefit of participating in the PREADVISE study is that early detection of memory changes can lead to early diagnosis and treatment. Also, some participants may decrease their risk of getting AD if the supplements are effective. The findings of this study may also help in the research and understanding of AD.

Only participants who are taking part in the SELECT study (a study that looks at the use of vitamin E and selenium for preventing prostate cancer) may apply to participate in the PREADVISE study about how useful vitamin E and selenium might be for preventing memory changes with age (including Alzheimer's disease and other disease that can affect the brain). African American and Hispanic men who are age 60 or older may take part. Men of other ethnic groups aged 62 or older may take part. The SELECT doctors or staff will review the applicant's medical history and drugs to verify that they have no conditions that would exclude them from this study. About 10,000 men will take part in this study.

The PREADVISE study examinations will be done during the participant's annual SELECT visit at the clinic where the SELECT studies are being conducted. There will be one study visit for each year the participants are in SELECT (7 to 12 visits). Each visit for PREADVISE will consist of a brief screening of the participant's memory, and an update (if any) of the participant's family history of dementia and medications. If memory changes are suggested by the brief memory screen, the participant will be asked to take a longer memory screen to further evaluate the potential for memory changes. If the longer memory screen also suggests problems with the participant's memory, the participant will be asked to see his family doctor or a PREADVISE doctor for a more complete medical exam to find the possible causes of the memory change. Results of the doctor's medical exam, with the consent of the participant, will be sent to the PREADVISE doctors for their review to help with the diagnosis. Results of the memory checks will not be given to the participants. However, if the participant does have a medical workup for memory changes, this information will be given to the family doctor after the medical workup is completed. A portion of the blood sample that was taken when the participant entered SELECT might be analyzed and tested for a genetic risk factor associated with Alzheimer's disease, called Apolipoprotein E (ApoE). The results of this test will be used for research purposes only.

ELIGIBILITY:
Inclusion Criteria:

* Participating in SELECT Prevention study;
* 62 years or older if other ethnic origin, or 60 years or older if African-American or Hispanic;
* General good health with no neurological or psychiatric illness.

Exclusion Criteria:

The SELECT doctors or staff will review the PREADVISE applicants' medical history and drugs to verify that they have no condition(s) that would exclude them from this study. The participant must not have any of the following neurological conditions based on self report (were told by a physician):

* Alzheimer's disease, or any other form of dementia such as Pick's disease, dementia with Lewy bodies, frontotemporal dementia, vascular dementia, significant cognitive and motor impairment from a stroke or corticobasal degeneration;
* Huntington's disease, epilepsy, Parkinson's disease, brain tumor, multiple sclerosis, manic-depressive disorder, or schizophrenia;
* The participant must not have had a head injury with prolonged loss of consciousness (over 30 minutes) within the past five years;
* The participant must not have a current alcohol or substance abuse diagnosis, or must have been treatment free for the past 24 months;
* The participant must not have had a diagnosis of depression or anxiety disorder in the past 4 months and must not currently be under treatment for depression or anxiety disorder. [A participant who was previously diagnosed with depression or anxiety disorder but completed treatment more than four months ago is eligible.];
* The participant must not currently use of any of the following medications: Aricept, Cognex, Exelon, Reminyl, or Hydergine;
* The participant must not have blindness, deafness, language difficulties or any other disability that may prevent completion of the memory screen.

Ages: 60 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participant will be recruited from primary care office visits
Sampling Method: Probability Sample
Enrollment: 4246 (Actual)
Dates: Start 2002-05 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
incidence of dementia (including Alzheimer's disease) | 7 to 12 years (depending on enrollment date)
  Participants will complete a modified Telephone Interview of Cognitive Status (TIC-S) to evaluate the onset of dementia

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Schmitt, PhD, Principal Investigator — Sanders-Brown Center on Aging; Richard Kryscio, PhD, Principal Investigator — Sanders-Brown Center on Aging
Locations (91):
- United States (84):
  - University of Alabama at Birmingham Preventive Medicine, Birmingham, Alabama
  - Alaska Regional Hospital, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University of California, San Diego - Chula Vista, Chula Vista, California
  - Glendale Memorial Hospital, Glendale, California
  - University of California, San Diego, La Jolla, California
  - VA Medical Center, Loma Linda, California
  - VAMC Long Beach, Long Beach, California
  - Northridge Hospital Medical Center, Northridge, California
  - Santa Rosa Memorial Hospital Regional CCOP, Santa Rosa, California
  - LABIOMED (Los Angeles Biomedical) Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Lionel B. Katchem, Upland, California
  - Rocky Mountain CC/Poudre Valley Hospital, Fort Collins, Colorado
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - DC United MBCCOP, Washington D.C., District of Columbia
  - Baptist Medical Center, Jacksonville, Florida
  - Kaiser Southeast Permanente Medical Group, Tucker, Georgia
  - Bliss Cancer Center/McFarland Clinic/Mary Greely MC, Ames, Iowa
  - Cedar Rapids CCOP, Cedar Rapids, Iowa
  - Genesis Medical Center, Davenport, Iowa
  - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Stormont-Vail Health Care/Cotton O'Neil Clinic, Topeka, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Our Lady of Bellefonte Hospital Inc., Ashland, Kentucky
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Louisville VA Medical Center, Louisville, Kentucky
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Berkshire Hematology Oncology/Bershire Medical Center, Pittsfield, Massachusetts
  - Bixby Oncology Center, Adrian, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Grand Rapids Clinical Oncology Program CCOP, Grand Rapids, Michigan
  - Monroe Clinic, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Duluth CCOP, Duluth, Minnesota
  - St. John's Regional Medical Center, Joplin, Missouri
  - St. John's Health System, Springfield, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Benefis Health Care, Great Falls, Montana
  - Good Samaritan Health Systems - Cancer Center, Kearney, Nebraska
  - Cancer Resource Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Missouri Valley Cancer Cons CCOP/Creighton University, Omaha, Nebraska
  - Washoe Medical Center, Reno, Nevada
  - VAMC New Jersey Health Care System, East Orange, New Jersey
  - Warren Hospital, Phillipsburg, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - Stratton Veterans Affairs Medical Center, Albany, New York
  - Bassett Research Institute, Cooperstown, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - NW Ohio Oncology Center/St. Luke's Hospital, Maumee, Ohio
  - St. Charles Hospital, Oregon, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Medical Center, Toledo, Ohio
  - Toledo CCOP, Toledo, Ohio
  - Toledo Clinic Inc., Toledo, Ohio
  - Muskogee Regional Medical Center, Muskogee, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital and Health Network, Bethlehem, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - York Cancer Center/Wellspan Health, York, Pennsylvania
  - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Baptist Memorial Hospital - Memphis, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Methodist Regional Cancer Center, Oak Ridge, Tennessee
  - Methodist Hospitals of Dallas, Dallas, Texas
  - Scott & White CCOP, Temple, Texas
  - Cascadia Clinical Trials at St. Joseph Hospital, Bellingham, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Northwest Hospital, Seattle, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
  - Sinai Samaritan Medical Center, Milwaukee, Wisconsin
- Ottawa General Hospital, Ottawa, Ontario, Canada
- Puerto Rico (6):
  - San Juan Dr. I. Gonzalez Martinez/Centro Medico, San Juan
  - Altamira Family Medicine, San Juan
  - Centro Clinico San Patricio, San Juan
  - Miguel Sosa Padilla, MD/San Juan City Hospital, San Juan
  - VAMC San Juan, San Juan
  - San Juan City Hospital - PR, Hematology Oncology Office, San Juan

REFERENCES:
- [Background] Lovell MA, Ehmann WD, Butler SM, Markesbery WR. Elevated thiobarbituric acid-reactive substances and antioxidant enzyme activity in the brain in Alzheimer's disease. Neurology. 1995 Aug;45(8):1594-601. doi: 10.1212/wnl.45.8.1594. PMID 7644059
- [Background] Sano M, Ernesto C, Thomas RG, Klauber MR, Schafer K, Grundman M, Woodbury P, Growdon J, Cotman CW, Pfeiffer E, Schneider LS, Thal LJ. A controlled trial of selegiline, alpha-tocopherol, or both as treatment for Alzheimer's disease. The Alzheimer's Disease Cooperative Study. N Engl J Med. 1997 Apr 24;336(17):1216-22. doi: 10.1056/NEJM199704243361704. PMID 9110909
- [Background] Markesbery WR, Carney JM. Oxidative alterations in Alzheimer's disease. Brain Pathol. 1999 Jan;9(1):133-46. doi: 10.1111/j.1750-3639.1999.tb00215.x. PMID 9989456
- [Background] Goodman PJ, Tangen CM, Darke AK, Arnold KB, Hartline J, Yee M, Anderson K, Caban-Holt A, Christen WG, Cassano PA, Lance P, Klein EA, Crowley JJ, Minasian LM, Meyskens FL. Opportunities and challenges in incorporating ancillary studies into a cancer prevention randomized clinical trial. Trials. 2016 Aug 12;17:400. doi: 10.1186/s13063-016-1524-9. PMID 27519183
- [Background] Mathews M, Abner E, Caban-Holt A, Dennis BC, Kryscio R, Schmitt F. Quality of education and memory test performance in older men: the New York University Paragraph Recall Test normative data. Curr Alzheimer Res. 2013 Sep;10(7):776-83. doi: 10.2174/15672050113109990140. PMID 23906000
- [Background] Kryscio RJ, Abner EL, Schmitt FA, Goodman PJ, Mendiondo M, Caban-Holt A, Dennis BC, Mathews M, Klein EA, Crowley JJ; SELECT Investigators. A randomized controlled Alzheimer's disease prevention trial's evolution into an exposure trial: the PREADViSE Trial. J Nutr Health Aging. 2013 Jan;17(1):72-5. doi: 10.1007/s12603-012-0083-3. PMID 23299383
- [Background] Abner EL, Dennis BC, Mathews MJ, Mendiondo MS, Caban-Holt A, Kryscio RJ, Schmitt FA; PREADViSE Investigators; Crowley JJ; SELECT Investigators. Practice effects in a longitudinal, multi-center Alzheimer's disease prevention clinical trial. Trials. 2012 Nov 20;13:217. doi: 10.1186/1745-6215-13-217. PMID 23171483
- [Background] Caban-Holt A, Abner E, Kryscio RJ, Crowley JJ, Schmitt FA. Age-expanded normative data for the Ruff 2&7 Selective Attention Test: evaluating cognition in older males. Clin Neuropsychol. 2012;26(5):751-68. doi: 10.1080/13854046.2012.690451. Epub 2012 May 31. PMID 22651854
- [Result] Ding X, Kryscio RJ, Turner J, Jicha GA, Cooper G, Caban-Holt A, Schmitt FA, Abner EL. Self-Reported Sleep Apnea and Dementia Risk: Findings from the Prevention of Alzheimer's Disease with Vitamin E and Selenium Trial. J Am Geriatr Soc. 2016 Dec;64(12):2472-2478. doi: 10.1111/jgs.14393. Epub 2016 Nov 1. PMID 27801937
- [Result] Abner EL, Kryscio RJ, Caban-Holt AM, Schmitt FA. Baseline subjective memory complaints associate with increased risk of incident dementia: the PREADVISE trial. J Prev Alzheimers Dis. 2015 Mar;2(1):11-16. doi: 10.14283/jpad.2015.37. PMID 26180776
- [Result] Kryscio RJ, Abner EL, Caban-Holt A, Lovell M, Goodman P, Darke AK, Yee M, Crowley J, Schmitt FA. Association of Antioxidant Supplement Use and Dementia in the Prevention of Alzheimer's Disease by Vitamin E and Selenium Trial (PREADViSE). JAMA Neurol. 2017 May 1;74(5):567-573. doi: 10.1001/jamaneurol.2016.5778. PMID 28319243
- [Derived] Ding X, Abner EL, Schmitt FA, Crowley J, Goodman P, Kryscio RJ. Mental Component Score (MCS) from Health-Related Quality of Life Predicts Incidence of Dementia in U.S. Males. J Prev Alzheimers Dis. 2021;8(2):169-174. doi: 10.14283/jpad.2020.50. PMID 33569563
- See also: Clinicaltrials.gov SELECT trial record — http://clinicaltrials.gov/show/NCT00006392
- See also: Southwest Oncology Group — http://www.swog.org